CLINICAL TRIAL: NCT00543491
Title: MK0767 and Sulfonylurea Combination Study (0767-027)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0767-027; 2007_629; MK-0767-027
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — MK0767

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0767

SUMMARY:
This study will assess MK0767's ability vs. placebo to control blood glucose in patients with type 2 diabetes and to gauge whether fasting blood glucose is lowered, blood fats are improved, and insulin levels are impacted.

This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes with inadequate glycemic control
* On Sulfonylurea monotherapy
* Male or non-pregnant Females
* Age 21 to 78 years, inclusive
* On a stable dose of sulfonylurea for at least 2 weeks prior to Visit 2/Week-6

Exclusion Criteria:

* History of Type 1 diabetes
* Patient is currently on insulin (monotherapy or in combination with oral agent), Rosiglitazone or pioglitazone or other PPAR-y agonists, Metformin agents
* Patients with history of or intolerance of PPAR-y agonists

Ages: 21 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2003-05; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC